CLINICAL TRIAL: NCT03362736
Title: An Early Access Program for Ustekinumab in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: An Early Access Program For Ustekinumab In Participants With Moderately To Severely Active Crohn's Disease
Status: No longer available | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108395; CNTO1275CRD3006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-11-30; First posted 2017-12-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — All participants will receive a single intravenous (IV) tiered dose of ustekinumab based on body weight at Week 0 (participants less than or equal to [<=] 55 kilogram [kg] will receive 260 milligram [mg] ustekinumab; > 55 kg to <= 85 kg will receive 390 mg ustekinumab; and > 85 kg will receive 520 mg ustekinumab infusion) during induction period. After the IV induction dose, all participants will receive the first maintenance dose of 90 mg ustekinumab subcutaneous (SC) injection 8 weeks later (Week 8). The participants with adequate response based on the physician's judgement will be subsequently treated with 90 mg ustekinumab SC injection with every 12 weeks through Week 80 and participants with an inadequate response to ustekinumab dosing every 12 weeks based on the physician's judgement will be subsequently treated with 90 mg of ustekinumab every 8 weeks through Week 80.
  Other Names: CNTO1275

SUMMARY:
The purpose of this program is to provide early access to ustekinumab where it is commercially unavailable for the treatment of participants with moderately to severely active Crohn's disease who have failed treatment with conventional Crohn's disease therapy (example, immunomodulators or corticosteroids) and Tumor Necrosis Factor alpha (TNF alpha) antagonist therapy (e.g., infliximab, adalimumab, certolizumab pegol, or their biosimilars), or who are intolerant to, or have a contraindication to these treatments. During the course of this early access program (EAP), through the reporting of serious adverse events (SAEs) and non-serious adverse drug reactions (ADRs) by participating physicians, information on the safety and tolerability of ustekinumab will be captured.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease or fistulizing Crohn's disease of at least three months' duration at the time of screening, with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Have active Crohn's disease, defined as:

  1. Baseline Crohn's disease activity index (CDAI) score of >= 220, and
  2. At least one of the following: a.) Abnormal C-reactive protein (CRP) levels at screening (defined by the participating physician/institution), b.) Fecal calprotectin level greater than or equal to (>=) 250 milligram per kilogram (mg/kg) at screening, c.) Endoscopy with evidence of active Crohn's disease during the current disease flare (defined as ulcerations in the ileum and/or colon). The endoscopy must have occurred within six months prior to baseline, d.) Harvey Bradshaw index (HBI) >= 5
* Otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. If there are abnormalities, they must be consistent with the underlying illness in the program population. This determination must be recorded in the participant's source documents and initialed by the physician
* Have failed treatment with conventional therapy (example, immunomodulators or corticosteroids) and Tumor necrosis factor alpha (TNFalpha) antagonist therapy (example, infliximab, adalimumab, certolizumab pegol, or their biosimilars), or are intolerant to, or have a contraindication to these treatments. The failure of conventional or biological therapy is defined as being a participant who, in the opinion of the health care provider, have not responded adequately to the treatment (that is, primary non-responders), or who lost response or became intolerant over time to the treatment (that is, secondary non-responders) based on the physician's judgement. The failure of conventional or TNF alpha antagonist therapy is defined as being a participant who, in the opinion of the health care provider, did not respond adequately to the treatment (that is, primary non-responders), or who lost response or became intolerant over time to the treatment (that is, secondary non-responders) based on the physician's judgement
* Meet one of the following conditions: a). Participant is female: Not of childbearing potential or of childbearing potential and has a confirmed negative pregnancy test and will be sexually inactive or agrees to practice a highly effective method of birth control, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patches, intrauterine devices, double-barrier method (example, condoms, diaphragms, or cervical caps, with spermicidal foam, cream, or gel) during and after participation in the early access program (EAP). Male condom and female condom should not be used together (due to risk of failure with friction). These restrictions apply through 20 weeks after receiving the last dose of ustekinumab, b). Participant is male: either sexually inactive or agrees to practice a highly effective method of birth control, such as a condom with spermicide during and after participation in the EAP, and agrees not to donate sperm during and after ustekinumab treatment. These restrictions apply through 20 weeks after receiving the last dose of ustekinumab

Exclusion Criteria:

* Has complications of Crohn's disease such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery, and would possibly confound the ability to assess the safety of treatment with ustekinumab
* Has had any kind of bowel resection within six months or any other intra-abdominal surgery within three months prior to baseline
* Has evidence of current active infection, including untreated latent tuberculosis, or a nodule suspicious for lung malignancy on screening or any other available chest radiograph, unless definitively resolved surgically or by additional imaging and with source document confirmation
* Has or is suspected to have an undrained abscess
* Enrolled in a clinical program of ustekinumab treatment of Crohn's disease in Brazil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- Brazil (6):
  - Hospital Nossa Senhora Das Gracas, Curitiba
  - Endogastro Clínica de Gastroenterologia e Endoscopia Digestiva Lida, Juiz de Fora
  - Instituto do Aparelho Digestivo, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - Hospital Copa D'Or, Rio de Janeiro

REFERENCES:
- See also: AN EARLY ACCESS PROGRAM FOR USTEKINUMAB IN PATIENTS WITH MODERATLY TO SEVERELY ACTIVE CROHN'S DISEASE — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR108395&attachmentIdentifier=abfcd363-8221-4ae8-a1d6-a37ca82615a5&fileName=CR108395_CSR_Synopsis.pdf&versionIdentifier=